CLINICAL TRIAL: NCT05536557
Title: Ultrasound-guided Bilateral External Oblique İntercostal (EOI) Plane Block in Patients Undergoing Laparoscopic Cholecystectomy: a Randomized Controlled Trial
Brief Title: Bilateral External Oblique İntercostal (EOI) Plane Block in Patients Undergoing Laparoscopic Cholecystectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, muhammet korkusuz, Principal Investigator, MD, Karaman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2022/11
Record Dates: First submitted 2022-09-06; First posted 2022-09-13 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; Acute Postoperative Pain; Nerve block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: There are two group;
  1. Experimental Group: Group (EOI) Plane Block ; A block needle will inserted with in-plane technique and 25 ml 0.25 bupivacaine will be applied to EOI plane. The same procedure will be repeated on the contralateral side. Patients will receive standard multimodal analgesia comprising paracetamol, deksketoprofen, and tramadol.
  2. Sham Comparator Group:The patients will not receive any intervention. Patients will receive standard multimodal analgesia comprising paracetamol, deksketoprofen, and tramadol.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator) Blocks will be administered after induction of general Anesthesia so participants will be blinded to which intervention they have had.Study investigators will not be aware of what group the participant belongs to when assessing the patient at post-operative period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (EOI) Plane Block (Active Comparator): After tracheal intubation, a high-frequency linear probe will be in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle identified at the level ribs 6 and 7 in line. A block needle will inserted with in-plane technique and 25 ml 0.25 bupivacaine will be applied to EOI plane. The same procedure will be repeated on the contralateral side. Patients will receive standard multimodal analgesia comprising paracetamol, deksketoprofen, and tramadol.
  Interventions: Other: Bilateral External Oblique İntercostal (EOI) Plane Block
- Group N (Sham Comparator): The patients in Group N will not receive any intervention. In the intervention and control groups, block sites will be covered with dressings, and patients and other health care workers will be blinded to treatment allocation. Patients will receive standard multimodal analgesia comprising paracetamol, deksketoprofen, and tramadol.
  Interventions: Other: Standard perioperative and postoperative multimodal analgesia

INTERVENTIONS:
Other: Bilateral External Oblique İntercostal (EOI) Plane Block — External Oblique İntercostal (EOI) Plane Block will be provided for postoperative pain for Laparoscopic Cholecystectomy with Bupivacaine. And patients will receive standard multimodal analgesia comprising paracetamol, deksketoprofen, and tramadol.
  Other Names: Quality of Recovery-15 score; Standard Pain Followup and Monitorization
  Arms: Group (EOI) Plane Block
Other: Standard perioperative and postoperative multimodal analgesia — Patients will receive standard multimodal analgesia comprising paracetamol, deksketoprofen, and tramadol for Laparoscopic Cholecystectomy.
  Other Names: Quality of Recovery-15 score; Standard Pain Followup and Monitorization
  Arms: Group N

SUMMARY:
This study will define the postoperative analgesic effect of ultrasound-guided bilateral External Oblique İntercostal (EOI) Plane Block and compare the control group in patients undergoing laparoscopic cholecystectomy.

The aim of this study is to compare postoperative opioid consumption of EOI plane block versus control group. It is hypothesized that postoperative opioid use will be less in patients with EOI plane block than in patients who only receive routine multimodal analgesia.

DETAILED DESCRIPTION:
Laparoscopy is a minimally invasive procedure, but postoperative pain is still the most common symptom after laparoscopic cholecystectomy (LC). Regional blocks used in addition to multimodal analgesia for postoperative pain after LC usually block the anterior branches of the intercostal nerves. After it was suggested by Hamilton et al. in 2018 that it could block the lateral cutaneous branches between T7-T11 intercostal nerve by administering local anesthetic to the thoracic facial plane and could be used in lateral abdominal surgeries, the EOI plane block has become a block that can be used for analgesic purposes in upper and lateral abdominal surgeries. Blocking the anterior and lateral branches together may produce analgesia in a wider area, resulting in less postoperative opioid consumption.

This study will be conducted as a single-center, prospective, randomized trial in a university hospital. Patients scheduled for elective laparoscopic cholecystectomy will be screened for enrollment in the study. After randomization, EOI Plane Block will be performed under ultrasound guidance after administering general anesthesia and prior to the skin incision. An anesthesiologist who performed blocks will not involve in the data collection. Other health care workers who will involve in the evaluation of postoperative opioid consumption,pain scores, nausea and vomiting, antiemetic use, and Quality of Recovery score will be blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

Patients' age between 18 and 70 years with American Society of Anesthesiology (ASA) physical status I-II, who will be scheduled for an elective laparoscopic cholecystectomy surgery included in the study.

Exclusion Criteria:

* presence of coagulation disorder
* infection at the injection site of the block
* known allergy to local anesthetics
* advanced hepatic or renal failure
* can not communicate in Turkish
* history of abdominal surgery or trauma
* conversion of laparoscopic to open surgery
* consumption of any pain killers within the 24 h before the operation
* chronic opioid consumption
* pregnancy
* alcohol or drug abuse
* body mass index (BMI) ≥ 35 kg m-2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Postoperative 24 hours
  If NRS score of the patient is equal or over 4, IV 50 mg tramadol will be applied as a rescue analgesic.

SECONDARY OUTCOMES:
Numerical Rating Scale scores | Postoperative 24 hours
  The primary outcome variable is Numerical Rating Scale scores both at rest and motion. A blinded anesthesiologist will assess postoperative pain during rest and motion at the postoperative 15th,30th and 60th minute, second,6th, 12th and 24th hour by using 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable).
Time to first rescue analgesic | Postoperative 24 hours
  The time for administration of first rescue analgesic.
Adverse events | Postoperative 24 hours
  Incidence of nausea and vomiting during postoperative 24 hour time period will be noted.
Metoclopromide consumption | Postoperative 24 hours
  The severity of the nausea will be assessed on a 4 -point scale (0=none 1=mild, 2=moderate 3=severe). If the patients nausea score is ≥2 the patient will receive 10 mg metoclopromide.
Sedation score | Postoperative 24 hour
  Sedation level of the patients will be assessed on a 4-point scale (0=alert, 1=sleepy, easy to arouse verbally, 2= drowsy, 3=does not open eyes to verbal commands) at postoperative 15th,30th and 60th minute, second, 6th, 12th and 24th hour.
Quality of recovery levels between groups by using QoR-15 questionnaire | Postoperative 24th hour
  A 15-parameter Quality of Recovery score (QoR-15) has been recommended as the optimum tool to evaluate overall patient-centers measures of recovery after surgery, including pain. It is a questionnaire that is given to patients to do postoperatively and is scored from 0 to 150 where 150 indicates that the patient has had an excellent recovery QoR-15 score will be recorded on the morning of operation and at the postoperative 24th hour.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Korkusuz, MD, Study Chair — Karaman Training and Research Hospital
Locations (1):
- Karaman Taining and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korkusuz M, Basaran B, Et T, Bilge A, Yarimoglu R, Yildirim H. Bilateral external oblique intercostal plane block (EOIPB) in patients undergoing laparoscopic cholecystectomy: A randomized controlled trial. Saudi Med J. 2023 Oct;44(10):1037-1046. doi: 10.15537/smj.2023.44.10.20230350. PMID 37777270